CLINICAL TRIAL: NCT03518190
Title: Early Detection of Pressure Induced Tissue Damage by Infrared Spectroscopy (ODP) Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yehuda Ullmann MD, Head of Plastic Surgery Department, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0039-18-RMB
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Pressure Ulcer Not Visible

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected pressure injury (Experimental): Patients evaluated with high-risk for pressure injury
  Interventions: Device: Infrared spectroscopy (ODP)

INTERVENTIONS:
Device: Infrared spectroscopy (ODP) — Infrared spectroscopy device will be used to detect non-visible pressure injuries

SUMMARY:
The aim of this study is to demonstrate that infrared spectroscopy is able to detect pressure injuries at a very early stage

DETAILED DESCRIPTION:
During pressure injuries formation early sub dermal bio signal appear. By applying infrared spectroscopy at a suspicions injury site on the human body and obtaining a reflected infrared light infrared allows to determine early formation of a pressure injury/

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 1 pressure injury
* Patients with high risk of developing pressure injury

Exclusion Criteria:

* Patients with stage 2 pressure injury or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Early detection of pressure induced tissue damage | Ten minutes
  Infrared spectroscopy will indicate on a system-defined scale (yes/no) whether or not the subject has a pressure injury
Pressure injury probability | Ten minutes
  Infrared spectroscopy will calculate using accepted statistical tools the probability of the subject getting a pressure injury within the next few days

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam healrh care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No